CLINICAL TRIAL: NCT03404752
Title: A Randomized, Multicenter Clinical Trial to Determine the Efficacy, Safety and Tolerability of Peg-filgrastim (Gema) Compared to Peg-filgrastim (Roche) for Prevention of Chemotherapy Induced Neutropenia in Patients With Breast Cancer
Brief Title: Pegfilgrastim-gema Compared to Pegfilgrastim-roche for Prevention of Induced Neutropenia in Breast Cancer Patients.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gema Biotech S.A. (Industry)
Collaborators: QUID Quality in Drugs and Devices Latin American Consulting SRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GEMPEGFIL001
Record Dates: First submitted 2016-02-15; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; Neutropenia; Peg-filgrastim; biosimilar
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peg-Neutropine® (Experimental): Study drug will be administered more than 24 hours after completion of chemotherapy and every 3 weeks with chemotherapy. Eligible patients scheduled to receive four or six cycles of chemotherapy in every three weeks will be screened in the preceding 28± 3 days and will be randomized (1:1) to one of two treatment arms (Peg-Filgrastim of GEMABIOTECH, or Peg-Filgrastim of Roche).
  Interventions: Drug: Peg-Filgrastim
- Neulastim® (Active Comparator): Study drug will be administered more than 24 hours after completion of chemotherapy and every 3 weeks with chemotherapy. Eligible patients scheduled to receive four or six cycles of chemotherapy in every three weeks will be screened in the preceding 28± 3 days and will be randomized (1:1) to one of two treatment arms (Peg-Filgrastim of GEMABIOTECH, or Peg-Filgrastim of Roche).
  Interventions: Drug: Peg-Filgrastim

INTERVENTIONS:
Drug: Peg-Filgrastim
  Other Names: Peg-Neutropine®; Neulastim®

SUMMARY:
This is a randomized, multicentre, Phase 3 study. Patients will be randomly assigned to the Study drug or its comparator. The study will be blinded for the staff members in charge of the endpoint assessment.

DETAILED DESCRIPTION:
Eligible patients will be scheduled to receive a chemotherapy regimen with risk of febrile neutropenia ≥20%. Study drug will be administered more than 24 hours after completion of chemotherapy and every 3 weeks with chemotherapy. Eligible patients scheduled to receive four or six cycles of chemotherapy in every three weeks will be screened in the preceding 28± 3 days and will be randomized (1:1) to one of two treatment arms (Peg-Filgrastim of GEMA BIOTECH, or Peg-Filgrastim of Roche).

A total of 4 or 6 cycles of chemotherapy supported by Peg-Filgrastim will be administered with an interval of three weeks between each cycle.

Patients will be followed up for 28± 3 days after the last dose of Peg-Filgrastim.

Hematological assessment (Absolute Neutrophil Count [ANC]) will be assessed on day 1 or up to -3 (before administration of anticancer chemotherapy), day 2 or 3 and 5 through 9 of the first cycle, and thereafter every day until post-nadir ANC recovery to ≥ 1.5 x 109/l following each cycle of chemotherapy. In the following cycles, hematological assessment shall be performed on day 1 or up to -3 (before administration of anticancer chemotherapy), on day 2 or 3 and on days 5 and 7. This schedule only applies if the subject did not develop Severe Neutropenia on the previous cycle. If the patient develops Severe Neutropenia on the first cycle or at any cycle, then the schedule corresponding to first cycle shall be followed.

During baseline (before the administration of Peg-Filgrastim), day 5 and day 9 following the first cycle of chemotherapy CD34+ (cluster of differentiation) count will be determined.

The study consists of:

* Screening (up to 4 weeks)
* Treatment period (6 cycles each of 3 weeks. i.e. a total of 18 weeks)
* Follow up period for safety (4 weeks after Peg-Filgrastim last dose)

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 70 years old.
* Patients diagnosed having high risk stage 2 or stage 3 or 4 of breast cancer (by histopathological or cytological diagnosis) and need neoadjuvant, adjuvant chemotherapy, or with metastatic disease.
* A priori has been decided to be treated with Peg-Filgrastim and subjects eligible for Peg-Filgrastim therapy according to indications and clinical use in the product monograph
* Patients scheduled to receive 4 or 6 cycles of chemotherapy (Taxane combinations) with prophylactic Peg-Filgrastim at 3 weeks interval. Monoclonal Antibodies in addition to Taxane regimens are permitted.
* Any acute adverse effects of prior therapy must have resolved to ≤ NCI CTCAE (Version 4.0) grade 1 (excluding alopecia) prior to Day 1 of Cycle 1
* Eastern Cooperative Oncology Group - ECOG Performance Status 0, 1 or 2 as determined on Day 1 or up to -3 of Cycle 1 prior to administration of chemotherapy
* Patients must have adequate organ function including the following:

  1. Adequate bone marrow functions, as determined within 3 days prior to administration of chemotherapy on Day 1 of Cycle 1 and as indicated by Hb ≥9,5 g/dl (transfusion permitted to be included in the trial ),WBC (white blood cell) ≥3,5 x 109/l, Absolute neutrophil count (ANC) ≥1.5 x 109/l, Platelets ≥95 x 109/l;
  2. Adequate renal and hepatic function, as determined within 3 days prior to administration of chemotherapy on Day 1 of Cycle 1 and defined as follows,

     1. Hepatic: Bilirubin ≤ 1.5 x the upper limit of normal (ULN) (unless elevation is known to be due to Gilbert's disease), Subjects must also meet one of the following criteria:

        1. Alkaline phosphatase within normal reference range and both AST (aspartate aminotransferase) and ALT (alanine aminotransferase) >2.5 x ULN; or
        2. Alkaline phosphatase <2.5 x ULN and both AST and ALT <1.5 x ULN; or
        3. Alkaline phosphatase <5 x ULN and both AST and ALT within normal reference range;
     2. Renal: Serum creatinine ≤ 1.5 mg/dl or creatinine clearance ≤ 60 ml/min (calculated according to the Cockcroft and Gault formula)
* Patients of child-bearing potential must have a negative pregnancy test within 3 days prior to the first dose of chemotherapy and at day 1 or up to -3 days of each Cycle) and use at least one form of contraception as approved by the investigator during the study.
* Life expectancy >6 months

Exclusion Criteria:

Safety of treatment dependent criteria:

* Presence of any serious concomitant systemic disorders incompatible with the administration of filgrastim, Peg-Filgrastim or any systemic disease that can influence the patient's safety according to doctor's diagnosis.
* History of hypersensitivity to Peg-Filgrastim, filgrastim or E.coli derived proteins.
* Serious local infection or active systemic infection within 10 days prior to enrollment or patients who have taken antibiotics within the previous 10 days
* Pregnant or breast-feeding patients
* Cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease (NYHA III or IV)
* Known bleeding disorder
* Patient known to have HIV, Hepatitis B, Hepatitis C or who have a positive serology for HIV, Hepatitis B or Hepatitis C at screening
* History or presence of sickle cell disease
* Concurrent or prior radiotherapy within four weeks of randomization

Criteria dependent on compliance with study procedures, or the evaluation of the response:

* Unwilling to use a reliable and acceptable contraceptive method throughout the study period (fertile patients only)
* Treatment with certain other agents to treat the malignant disease
* Known drug addiction, including alcoholism
* Treatment with any investigational product within 30 days prior to study drug administration
* Concurrent prophylactic antibiotics
* Previous participation in this study.
* Already involved in another trial.
* History of bone marrow or stem cell transplantation.
* Previous therapy should not have included G-CSF (granulocyte-colony stimulating factor)

Previous participation in this study: Subjects who are considered screening failures are allowed to be re-screened, except if have started chemotherapy. In case of re-screening the following assessments and evaluations do not have to be repeated: Demographics, Medical history, HIV, Hepatitis B and C serology.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Efficacy: Duration (in days) of severe neutropenia-DSN | Day 5 to day 9 of the first cycle
  ANC (Absolute Neutrophil Count) < 500/mm3 in the first cycle of chemotherapy.

SECONDARY OUTCOMES:
Clinical Efficacy: Incidence of severe neutropenia | Day 5 to Day 21 during 4 - 6 cycles
  ANC (Absolute Neutrophil Count) <500/mm3 or 0.5 x 109/l not associated with fever across the cycles
ANC nadir | Day 5 to Day 21 during 4 - 6 cycles
  Determination of ANC decreasing (depth of ANC nadir) and time to the post nadir ANC recovery (ANC ≥ 1500 /mm3)
Incidence of neutropenia | Day 5 to Day 21 during 4 - 6 cycles
  Incidence of Grade 3 neutropenia (ANC <1000 - 500/mm3) . incidence of Febrile Neutropenia-FN [defined as ANC <1000/mm3 or 1.0 x 109/l and a single temperature of >38.3° C (101° F) or a sustained temperature of ≥38° C (100.4° F)] for more than one hour by cycle and across the cycles. incidence of ANC <500/mm3 and body temperature of >38.3°C.
Fever | Day 5 to Day 21 during 4 - 6 cycles
  Incidence of fever (temperature of >38.3° C - 101° F)
infections | Day 5 to Day 21 during 4 - 6 cycles
  Incidence of infections
IV anti-infectives | Day 5 to Day 21 during 4 - 6 cycles
  Incidence of need for IV anti-infectives
Post-chemotherapy hospitalization | Day 5 to Day 21 during 4 - 6 cycles
  Incidence and duration of post-chemotherapy hospitalization
Hospitalization due to neutropenia | Day 5 to Day 21 during 4 - 6 cycles
  Incidence and duration of hospitalization as a result of neutropenia
Mortality | Day 5 to Day 21 during 4 - 6 cycles
  Mortality due to infection
Pharmacodynamics | Day 5 and 9 of the first cycle
  The mobilization of CD34+ cells
Incidence of Adverse Drug Reactions (safety and tolerability) as assessed by CTCAE v4.0 | Day 5 to Day 21 during 4 - 6 cycles
  Frequency of patients who withdraw the study drug due to lack of tolerance Frequency of patients who withdraw the study drug treatment due to any reason Incidence of local tolerability at the injection site
Immunogenicity | Day 5 and Day 28 of the last cycle
  Neutralizing Antibody (NABs) Titer and Binding Antibodies (BABs) to Peg-Filgrastim (anti-rG-CSF [Recombinant Granulocyte-Colony stimulating factors] antibodies greater or equal to a determined concentration expressed in U/mL) will be measured using validated methods

CONTACTS AND LOCATIONS:
Overall Officials: Ezequiel Klimovsky, MD, Study Chair — QUID quality in drugs and devices LATAM consulting SRL
Locations (1):
- COIBA, Buenos Aires, Bs As, Argentina

IPD SHARING:
Plan to Share IPD: Undecided